CLINICAL TRIAL: NCT05186532
Title: To What Extent Does Application of Dry Heat is Effective in Promoting Episiotomy Wound Healing and Reducing Pelvic Pain Among Primipara Women?
Brief Title: Dry Heat Versus Sitz Bath On Episiotomy Wound Heating And Pelvic Pain
Acronym: Dry_Heat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Zohour Ibrahim Mahmoud Rashwan, lecturer, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 4445566888
Record Dates: First submitted 2021-12-23; First posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Wound Heal; Pain, Postoperative
Keywords: Infrared Rays; Heat; Hydrotherapy; episiotomy; Pelvic Pain; wound healing
MeSH Terms: conditions — Pain, Postoperative; Pelvic Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry heat group (Experimental): infra red-light therapy that supplies radiant heat or infra-red rays to produce heat to the episiotomy wound.
  Interventions: Radiation: Dry Heat Application
- Moist heat group (Active Comparator): warm sitz bath in which a woman is asked to sit in a warm water tub up to the hip level.
  Interventions: Other: Moist Heat Application

INTERVENTIONS:
Radiation: Dry Heat Application — 50 postnatal women they were encouraged to place an infrared lamp at distance of 45 cm from the perineum and the heat produced with 230 volts for ten minutes. But the mother is checked after the first five minutes to make sure that she was not being burned. The researchers were demonstrated for each woman how to use infrared lamp, and it was followed by re demonstrations and discussions. After 12 hours of episiotomy this procedure was carried out in the morning and evening for ten consecutive days. The researcher gives the infrared lamp device for each woman then restore it after completion of the study.
  Arms: Dry heat group
Other: Moist Heat Application — included 50 postnatal women they were encouraged to sit in a basin (tub) of warm water (45 o C -59 o C) without pressure on the perineum and with the feet flat on the floor for 10 minutes. The researchers were demonstrated for each woman how to do warm sitz bath, and it was followed by re demonstrations and discussions. After 12 hours of episiotomy this procedure was carried out in the morning and evening for ten consecutive days.
  Arms: Moist heat group

SUMMARY:
Objective: To compare the effect of dry heat versus moist heat application on episiotomy wound healing and pain among postnatal mothers.

Research hypothesis H0: Postnatal mothers who apply dry heat on their episiotomy wound experience the same wound healing and pain as those who apply moist heat.

H1: Postnatal mothers who apply dry heat on their episiotomy wound experience faster wound healing and less pain than those who apply moist heat.

H2: Postnatal mothers who apply moist heat on their episiotomy wound experience faster wound healing and less pain than those who apply dry heat.

DETAILED DESCRIPTION:
A quasi-experimental study was carried out at Abu EL-Matamer Central Hospital and Housh Issa Central Hospital. A sample of 100 postnatal women were randomly assigned into two equal groups. Women in the control group received the moist heat, which entails; sitting in a warm water tub up to the hip level. While, the study group were subjected to infra red-light therapy that supplies radiant heat or infra-red rays to produce heat to the episiotomy wound.

Women who fulfilled the criteria from the postnatal inpatient ward at Abu EL-Matamer Central Hospital and Housh Issa Central Hospital in El-Beheira Governorate. Each woman was randomly assigned to one of the (dry heat or moist heat) groups. The researchers explained the aim of the study to every woman, and then her consent to participate in the study was obtained.

All study subjects were individually interviewed by the researchers on the first two hours after delivery during hospital stay to collect the basic data, episiotomy pain intensity was assessed by, as well as the researchers inspect the episiotomy site for Redness, Edema, Ecchymosis, Discharge and Approximation of the wound edges using REEDA scale within 2 hours after episiotomy repair to evaluate wound healing (Pretest).

After the assessment the researchers provided clear and concise information through illustrative pamphlet for the both groups.

Dry heat group included 50 postnatal women they were encouraged to place an infrared lamp at distance of 45 cm from the perineum and the heat produced with 230 volts for ten minutes. But the mother is checked after the first five minutes to make sure that she was not being burned. The researchers were demonstrated for each woman how to use infrared lamp, and it was followed by re demonstrations and discussions. After 12 hours of episiotomy this procedure was carried out in the morning and evening for ten consecutive days. The researcher gives the infrared lamp device for each woman then restore it after completion of the study.

Moist heat group included 50 postnatal women they were encouraged to sit in a basin (tub) of warm water (45 o C -59 o C) without pressure on the perineum and with the feet flat on the floor for 10 minutes. The researchers were demonstrated for each woman how to do warm sitz bath, and it was followed by re demonstrations and discussions. After 12 hours of episiotomy this procedure was carried out in the morning and evening for ten consecutive days.

At the end of the session the researchers gave each woman health education about the importance of follow-up to ensure woman compliance for the interventions they assigned to it and to assess wound healing. The researchers motivated the women to perform the interventions they assigned to it through daily telephone calls by reminding the women with its benefits and importance of follow up.

Follow up: Women of the two groups were instructed to come to the obstetric outpatient clinic at Abu EL-Matamer Central Hospital and Housh Issa Central Hospital for follow up visits during the morning shift on the 5th and 10th day post-partum, the perineal area was observed for redness, edema, ecchymosis, discharge and approximation of the skin as well as perineal pain. During each follow up visit the researchers had evaluated the episiotomy pain intensity using and episiotomy wound healing.

ELIGIBILITY:
Inclusion Criteria:

* Primipara
* First 2 hours after delivery
* Have a normal vaginal delivery
* Have episiotomy
* complaining of perineal discomfort (pain)
* Having a telephone for contact

Exclusion Criteria:

* The women who were
* use any pain-relieving drug
* labor complications
* postpartum complications
* diabetes
* anemia
* Illiterate

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — women with normal vaginal delivery and episiotomy and
Enrollment: 100 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Pelvic pain | After 10 days
  The researchers measured the pelvic pain intensity using Visual analogue scale: This scale was adopted and translated to an Arabic version to be used in the current study. It was developed by Melzack and Katz (1994). It is a self-reported device consisting of a horizontal line used for subjective estimation of patient's pain. It comprises 10-point numerical scale, corresponding to the degree of pain with zero representing no pain and 10 representing the worst degree of pain. Scores 1, 2, 3 indicate mild pain, while 4, 5, 6 scores indicate moderate pain and 7, 8, 9 scores indicate severe pain; finally, 10 indicate the worst unbearable pain
Episiotomy wound healing | After 10 days
  The researchers assessed episiotomy wound healing using The standardized Redness, Oedema, Ecchymosis, Discharge, Approximation (REEDA) scale ; The REEDA scale is an observational check list used for assessing perineal wound healing that was primarily developed by Davidson (1974). It can be used to assess all types of postpartum perineal trauma. It has five components namely Redness, Edema, Ecchymosis, Discharge and Approximation of the wound edges. Each component takes a score ranged from 0 to 3 . Total REEDA score ranges between 0 and 15. Higher score indicates poor wound healing while lower score indicates good wound healing. The total score of REEDA scale was categorized as follows; Completely healed from 0 to 2 , Moderately healed from 3 to 5 , Mildly healed from 6 to 8, and Not healed from 9 to 15

CONTACTS AND LOCATIONS:
Overall Officials: Eman m Taha, professor, Study Chair — Alexandria University
Locations (1):
- Faculty of Nursing, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Priddis H, Schmied V, Dahlen H. Women's experiences following severe perineal trauma: a qualitative study. BMC Womens Health. 2014 Feb 21;14(1):32. doi: 10.1186/1472-6874-14-32. PMID 24559056
- [Background] Steen M, Cummins B. How to alleviate perineal pain following an episiotomy. Nurs Stand. 2016 Mar 30;30(31):34-7. doi: 10.7748/ns.30.31.34.s43. No abstract available. PMID 27027195
- [Background] Swain J, Dahlen HG. Putting evidence into practice: a quality activity of proactive pain relief for postpartum perineal pain. Women Birth. 2013 Mar;26(1):65-70. doi: 10.1016/j.wombi.2012.03.004. Epub 2012 May 8. PMID 22575710
- [Background] Petersen MR. Review of interventions to relieve postpartum pain from perineal trauma. MCN Am J Matern Child Nurs. 2011 Jul-Aug;36(4):241-5. doi: 10.1097/NMC.0b013e3182182579. PMID 21709521
- [Background] Sarbaz Z, Yazdanpanahi Z, Hosseinkhani A, Nazari F, Akbarzadeh M. The Effect of Sitz Bath of Hydro-Alcoholic Extract of Myrrh Gum on Episiotomy Wound Healing in Nulliparous Women. J Family Reprod Health. 2019 Jun;13(2):89-97. PMID 31988645